CLINICAL TRIAL: NCT00981409
Title: Clinical Evaluation of GSK576428 (Fondaparinux Sodium) in the Treatment of Acute Pulmonary Thromboembolism (PE)
Brief Title: The Treatment of Acute Pulmonary Thromboembolism (PE) of GSK576428 (Fondaparinux Sodium) in Japanese Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106206
Record Dates: First submitted 2009-09-03; First posted 2009-09-22 (Estimated); Results first posted 2009-12-10 (Estimated); Last update posted 2016-12-16 (Estimated); Status verified 2016-11

CONDITIONS: Embolism, Pulmonary
Keywords: Fondaparinux sodium; contrast-enhanced MDCT; Deep Vein Thrombosis; Pulmonary thromboembolism
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — Fondaparinux; Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fondaparinux (Experimental)
  Interventions: Drug: Fondaparinux sodium
- unfractionated heparin (Other)
  Interventions: Drug: unfractionated heparin (UFH)

INTERVENTIONS:
Drug: Fondaparinux sodium — The dose of Fondaparinux will be determined based on a subject's body weight (<50 kg, 5 mg; 50 to 100 kg, 7.5 mg; >100 kg, 10 mg) and administered once daily by subcutaneous (SC) injection.
  Other Names: GSK576428
  Arms: Fondaparinux
Drug: unfractionated heparin (UFH) — UFH therapy will be started on Day 1 while adjusting activated partial thromboplastin time (aPTT) to maintain aPTT 1.5 to 2.5 times control.
  Arms: unfractionated heparin

SUMMARY:
The primary objective is to evaluate the efficacy (as measured by the rate of recurrent symptomatic Venous Thromboembolism [VTE] (i.e., Pulmonary thromboembolism [PE] and Deep Vein Thrombosis [DVT])) and safety of GSK576428 as the initial treatment in subjects with acute PE in an open-label design.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a confirmed diagnosis (by Multi detector-row CT [MDCT]) of acute symptomatic PE who are hemodynamically stable (i.e., the condition where anticoagulant therapy alone are indicated) (the time from onset should be no longer than 5 days, and subjects with or without symptomatic DVT are eligible)
* Age: >=20 years
* Gender: No restriction Female subjects must either be of non-childbearing potential (post-menopausal >1 year, hysterectomy, or sterilization), or of childbearing potential, has a negative pregnancy test at screening, and agree to use contraception throughout the study period.
* Hospitalization status: Subjects who are able to stay at the hospital at least during the initial treatment period.
* Written informed consent from the subject him/herself or his/her legally acceptable representative. Written informed consent from the subject's legally acceptable representative must be obtained if the subject is incapable of giving consent.

Exclusion Criteria:

* Shock or hemodynamic instability*.

  *: Defined as shock or decreased blood pressure (systolic blood pressure <90 mmHg or >=40 mmHg) lasting for at least 15 minutes and does not represent hemodynamically unstable conditions due to newly emergent arrhythmia, dehydration or sepsis.
* Right cardiac function failure detected by echocardiography at screening.
* Requirement for surgical thrombectomy, catheter intervention and thrombolytic therapy for the current PE.
* Subjects (for example, with free-floating thrombus in the femoral vein or ilium by MDCT at screening) for whom insertion of inferior vena cava filter is indicated or subjects in whom inferior vena cava filter is present.
* Prior to entry into the study, therapeutic dosage of anticoagulants for more than 24 hours to treat the current episode.
* Active, clinically significant bleeding
* Thrombocytopenia (platelet count <10×10⁴/µL at screening)
* Concurrent conditions with bleeding risk (e.g., ulcer of the gastrointestinal tract, diverticulitis of the gastrointestinal tract, colitis, acute bacterial endocarditis, severe hypertension*, or severe diabetes) or bleeding tendency.

  *: systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
* Severe hepatic disorder
* Known hypersensitivity to heparin, low-molecular-weight heparin (LMWH) or warfarin
* Previous history of cerebral hemorrhage
* Brain, spinal, or ophthalmological surgery within 3 months prior to entry into this study
* Previous history of Heparin-induced thrombocytopenia
* Patients for whom anticoagulant therapy is contraindicated or who cannot be taken off anticoagulant therapy due to coexistent condition (e.g. prosthetic heart valve implant).
* Severe renal disorder (serum creatinine >2.0 mg/dL [180 µmol/L] at screening) in a well hydrated subject
* Documented hypersensitivity to contrast media
* Use of any contraindicated drug that cannot be combined with the injection of contrast medium [e.g., antihyperglycemic metformin hydrochloride (Glycoran®, Melbin®)]
* Participation in any other therapeutic drug study or a clinical study within 6 months prior to entry into this study
* Previous participation in a study of GSK576428
* Drug or alcohol abuse
* Systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg
* Recent surgery within 3 days prior to entry into the study
* Life expectancy <3 months
* Pregnant women, nursing mothers, women who may be pregnant, or women contemplating pregnancy during the study period
* Others whom the investigator or subinvestigator considers not eligible for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (17):
- Japan (17):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Nakamura M, Okano Y, Minamiguchi H, Munemasa M, Sonoda M, Yamada N, Hanzawa K, Aoyagi N, Tsujimoto H, Sarai N, Nakajima H, Kunieda T. Multidetector-row computed tomography-based clinical assessment of fondaparinux for treatment of acute pulmonary embolism and acute deep vein thrombosis in Japanese patients. Circ J. 2011;75(6):1424-32. doi: 10.1253/circj.cj-10-1036. Epub 2011 Apr 22. PMID 21512258
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 106206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 106206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 106206 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Fondaparinux Sodium (FPX): The dose of FPX was determined based on a participant's body weight (<50 kg, 5 mg; 50 to 100 kg, 7.5 mg; >100 kg, 10 mg) and administered once daily by subcutaneous (SC) injection for 5-10 days as a general rule. Concomitant warfarin therapy (administered no later than 72 hours after the first dose of FPX) was continued up to Day 90 (±7) at a dose adjusted to maintain the prothrombin time international normalized ratio (PT-INR) between 1.5 and 3.0.
- Unfractionated Heparin (UFH): The dose of UFH was adjusted to maintain activated partial thromboplastin time (aPTT) at 1.5 to 2.5 times control and administered by intravenous (IV) drip bolus injection followed by IV infusion for 5-10 days as a general rule. Concomitant warfarin therapy (administered no later than 72 hours after the first dose of UFH) was continued up to Day 90 (±7) at a dose adjusted to maintain the PT-INR between 1.5 and 3.0.
Period: Overall Study
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Started | 30 | 11
Completed | 24 | 10
Not Completed | 6 | 1
Not completed — Adverse Event | 4 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Prostate Cancer Treatment before Trial | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH) | Total
Number analyzed (Participants) | 28 | 10 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] — Analysis population was Full Analysis Set (FAS); all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute pulmonary thromboembolism (PE).
  years | 68.5 (11.4) | 62.6 (14.1) | 67.0 (12.2)
Gender [Count of Participants; unit: Participants] — Analysis population was Full Analysis Set (FAS); all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute pulmonary thromboembolism (PE).
  Participants
    Female | 13 | 7 | 20
    Male | 15 | 3 | 18
Race/Ethnicity, Customized [Number; unit: participants] — Analysis population was Full Analysis Set (FAS); all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute pulmonary thromboembolism (PE).
  participants
    Asian-Japanese | 28 | 10 | 38
Body weight [Number; unit: kilograms (kg)] — Participants were weighed at screening (within 10 days before randomisation). Analysis population was Full Analysis Set (FAS); all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute pulmonary thromboembolism (PE).
  kilograms (kg)
    <50 kg | 5 | 1 | 6
    50-100 kg | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants With Recurrent or New Symptomatic Venous Thromboembolism (VTE)
Description: VTE (pulmonary thromboembolism [PE] and/or deep vein thromboembolism [DVT]) was adjudicated blindly by the Central Independent Adjudication Committee of Efficacy (CIACE).
Time Frame: From Day 1 to Day 90 (±7 days)
Population: Full Analysis Set (FAS): all participants receiving at least one dose of medication (FPX or UFH) who had efficacy data and had a confirmed diagnosis of acute pulmonary thromboembolism (PE)
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 10
percentage of participants | 0 | 0

2. Secondary Outcome: The Percentage of Participants With Recurrent or New Symptomatic/Asymptomatic Venous Thromboembolism (VTE) (by Type)
Description: as for outcome 1
Time Frame: From Day 1 to Day 90 (±7 days)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 10
percentage of participants
  Symptomatic DVT only | 0 | 0
  (Symptomatic) Non-fatal PE | 0 | 0
  (Symptomatic) Fatal PE | 0 | 0
  Asymptomatic DVT only | 0 | 0
  Asymptomatic PE | 0 | 0

3. Secondary Outcome: The Percentage of Participants With Perfusion Lung Scan Results Scored as Improved, no Change, or Worse
Description: "Improved," "No change," or "Worse" was adjudicated blindly by the Central Independent Adjudication Committee of Efficacy (CIACE). Each category is adjudicated by comparison with the perfusion score at baseline by the CIACE.
Time Frame: Baseline, Days 5-10 (the day when the medication [FPX or UFH] was finished /discontinued) (+/-1)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 10
percentage of participants
  Improved | 78.6 | 90.0
  No change | 21.4 | 10.0
  Worse | 0 | 0

4. Secondary Outcome: Total Perfusion Score at Baseline and Mean Change From Baseline at Days 5-10
Description: The perfusion score (0: no perfusion; 0.25, 0.5, 0.75, 1: normal) in each of the six lobes of the lung was adjudicated blindly by the Central Independent Adjudication Committee of Efficacy (CIACE). Total perfusion score (r) was calculated as: r = (0.25 x right lower lobe) + (0.12 x right middle lobe) + (0.18 x right upper lobe) + (0.20 x left lower lobe) + (0.12 x lingula) + (0.13 x left upper lobe).
Time Frame: Baseline, Days 5-10 (the day when the medication [FPX or UFH] was finished /discontinued) (+/-1)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 28 | 10
points on a scale
  Baseline | 0.654 (0.141) | 0.586 (0.237)
  Change from baseline, Days 5-10 (+/-1) | 0.101 (0.079) | 0.185 (0.148)

5. Secondary Outcome: The Percentage of Participants With a Bleeding Event
Description: Bleeding events (major bleeding [clinically overt bleeding with: fatality, location in critical organ, a fall in hemoglobin >=2 g/dL, or a transfusion >=2 units], minor bleeding [clinically overt bleeding and not adjudicated as major bleeding]) were adjudicated blindly by the Central Independent Adjudication Committee of Safety (CIACS).
Time Frame: FPX or UFH treatment period (Days 5-10, on average)
Population: Safety population: all participants who received at least one dose of medication (FPX or UFH).
Measure: Number; unit: percentage of participants
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Number analyzed (Participants) | 31 | 10
percentage of participants
  Major bleeding only | 0 | 0
  Minor bleeding | 9.7 | 0
  Any bleeding (major and/or minor bleeding) | 9.7 | 0

ADVERSE EVENTS:
Time Frame: FPX or UFH treatment period (Days 5-10 days, on average)
Description: SAEs and AEs were collected for the Safety Population (all participants who received at least one dose of medication [FPX or UFH]). One participant was randomized to UFH, but was incorrectly administered FPX.
Arm/Group | Fondaparinux Sodium (FPX) | Unfractionated Heparin (UFH)
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/10
Other Adverse Events (participants affected / at risk) | 17/31 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium (FPX) (N=31) | Unfractionated Heparin (UFH) (N=10)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fondaparinux Sodium (FPX) (N=31) | Unfractionated Heparin (UFH) (N=10)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 3 | 1
Urinary tract infection (Infections and infestations) | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Occult blood (Investigations) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Genital erosion (Reproductive system and breast disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.